CLINICAL TRIAL: NCT03621423
Title: The Use of Ultrasound for Botulinum Toxin Subscapularis Muscle Injection Guidance in Spastic Hemiplegic Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, Motti Ratmansky, MD, Director of the pain unit, Loewenstein Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0017-17-LOE
Record Dates: First submitted 2018-07-30; First posted 2018-08-08 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Hemiplegia, Spastic
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: Patient will be positioned lying on side with the hemiplegic side up. The shoulder will be placed in a flexion and external rotation/abduction position, as possible by the patient, to give the ultrasound probe access to the posterior axillary fold.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ultrasound guided injection — Patient will be positioned lying on side with the hemiplegic side up. The shoulder will be placed in a flexion and external rotation/abduction position, as possible by the patient, to give the ultrasound probe access to the posterior axillary fold.
  As previously described in the literature, a line of best fit was calculated by bisection of hypothetical line connecting the inferior spine and the acromial tip, an 18-gauge, 10-cm needle will be inserted under direct ultrasound guidance and by a nerve stimulation . After placing the needle tip in the target point's 100 units of botulinum toxin will be injected.

SUMMARY:
The aim of the study is to describe the efficacy of a new approach to the subscapularis muscle under US guidance for the injection of botulinum toxin in patients that underwent a stroke suffering from hemiplegic shoulder pain.

Pain and spastic shoulder are common findings in hemiplegic patients following a stroke.

The pain interferes with rehabilitation prolonging hospitalization and is related with decreased quality of life.

There is a close relationship between spasticity of the subscapularis muscle and pain The patients show a clinical picture of adduction and internal rotation of the shoulder, elbow and wrist and fingers flexion with a limited external rotation of the shoulder.

The investigators suggest that paralyzing the subscapularis muscle with botulinum toxin may alleviate pain in the hemiplegic shoulder. Best produced when injected in a specific area of the muscle where a higher concentration of motor points exists.

DETAILED DESCRIPTION:
Treatment using injection of botulinum toxin to the subscapularis spastic muscle has been described in the literature and is a common practice in hemiplegic shoulder. The Injection technic in this pathology is described by using anatomical landmarks of the shoulder region without using medical imaging.

On the other hand, injections to the subscapularis muscle has also been described using ultrasound guidance but not for this specific pathology.

There are no evidence-based guidelines describing us guided spastic subscapularis muscle injection. Injecting this muscle while in its spastic state requires a modulated approach Harrison et.al described cadaveric dissections of the subscapularis muscle and proposed a technique to reach the motor point zone of this muscle In our study the investigators follow the injection description published by Dong Wook Rha on cadavers based on Harrison's lateral approach description. The Ultrasound enables a correct identification of the target muscle avoiding possible complication of vessel or pulmonary puncture In our study the investigators will try to prove the efficacy of the lateral approach to the subscapularis muscle using ultrasound and nerve stimulator

ELIGIBILITY:
Inclusion Criteria:

Post stroke patients

* Complaints of pain in hemiplegic shoulder
* Spasticity of subscapularis muscle
* Coherent
* Hebrew speakers

Exclusion Criteria:

* Aphasia
* Allergy to botulinum toxin
* Pregnant women

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
The Modified Ashworth scale (MAS) | The MAS will be assessed twice: the first time before the injection and the second time, in order to assess change from baseline measure, two weeks following the injection
  measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity.
  * 0: No increase in muscle tone
  * 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  * 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  * 2: More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  * 3: Considerable increase in muscle tone, passive movement difficult
  * 4: Affected part(s) rigid in flexion or extension

SECONDARY OUTCOMES:
The Fugl-Meyer Assessment (FMA) | The FMA will be assessed twice: the first time before the injection and the second time two weeks following the injection
  a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
Visual Analogue Scale (VAS) | The VAS will be assessed twice: the first time before the injection and the second time two weeks following the injection
  a measurement instrument that tries to measure the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain (0-10). The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations.
The Brief Pain Inventory - Short Form (BPI-sf) | The BPI-sf will be assessed twice: the first time before the injection and the second time two weeks following the injection
  a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale.